CLINICAL TRIAL: NCT06935058
Title: Effectiveness of Chocolate Milk in Recovery Among Elite Kayakers: A Metabolic and Inflammatory Perspectives
Brief Title: Effectiveness of Chocolate Milk in Recovery Among Highly Trained Kayakers: A Metabolic and Inflammatory Perspectives
Acronym: Kayakers2025
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Anna Kasperska, PhD, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Kayakers 2025
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Inflammatory Responses; Muscle Fatigue; Recovery Time; Hunger
Keywords: insulin; kayakers; grelin; glucose; glycogen; regeneration; fatigue
MeSH Terms: conditions — Insulin Resistance; Fatigue | interventions — Water

STUDY DESIGN:
Intervention Model Description: Kayakers (both sexes), split into two groups:
  1. experimental group (n=15, 400 ml of chocolate milk),
  2. control group (n=15, 400 ml of water). Blood samples (capillary and venous) will be collected pre-exercise, post-exercise, and 1 hour post-consumption.
  All indicated parameters will be determined using the equipment of the biochemical laboratory of the University of Physical Education in Poznań, Branch in Gorzów Wielkopolski, and purchased commercial kits (immunoenzymatic ELISA tests). The analyses will be performed by the included project contractors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chocolade milk arm (Experimental): Participants will consume 400 ml of chocolate milk after exercise.
  Interventions: Other: Chocolade milk
- Control arm (Placebo Comparator): Participants will consume 400 ml of water after exercise.
  Interventions: Other: Water (Placebo)

INTERVENTIONS:
Other: Chocolade milk — Participants will drink 400 ml of chocolate milk after exercise.
  Arms: Chocolade milk arm
Other: Water (Placebo) — Participants will drink 400 ml of water after exercise.
  Arms: Control arm

SUMMARY:
Kayaking requires high energy expenditure and optimal metabolic adaptation for performance and recovery. While research on other sports exists, the effects of chocolate milk on kayakers' recovery remain unexplored.

Intensive kayaking induces physical stress, necessitating precise energy balance monitoring. This study evaluates metabolic and inflammatory markers, including glucose, glycogen, insulin, creatine kinase (CK), interleukin-6 (IL-6), ghrelin, leptin, peptide YY, peripheral blood morphology, and blood gas parameters to assess fatigue and recovery.

Chocolate milk, with its ideal carbohydrate-to-protein ratio, supports glycogen replenishment, muscle repair, hydration, and oxidative stress reduction. Studies suggest it may outperform commercial sports drinks in endurance recovery by limiting muscle damage, inflammation, and improving acid-base balance.

Findings will reveal whether chocolate milk enhances energy recovery, reduces muscle damage, and mitigates inflammation, contributing to endurance sports nutrition strategies

DETAILED DESCRIPTION:
Kayaking, as an endurance discipline, is associated with high energy expenditure and the need to optimize metabolic and hormonal processes in order to maximize efficiency and effective regeneration. Intense physical effort leads to significant changes in muscle metabolism and triggers an inflammatory response in the body. Such large loads require precise monitoring of energy balance and effective regeneration strategies. In the context of such intensive activity, monitoring biochemical indicators becomes crucial. They will allow for the assessment of the degree of fatigue and the course of regeneration processes. As part of the project, key metabolic and inflammatory indicators will be analyzed, such as glucose, glycogen and insulin levels, which will allow for the assessment of the efficiency of energy resource management. In addition, muscle damage indicators will be monitored, such as creatine kinase (CK) and interleukin 6 (IL-6), which will allow for the assessment of fatigue and regeneration processes in athletes.

Acid-base balance, a crucial factor in buffering lactic acid and oxygen transport to muscles, will be analyzed via blood gasometry (ABG). Lactic acid (LA) levels will also be monitored as a key fatigue indicator. Blood morphology analysis will complement the study, assessing the impact of intense exercise and recovery strategies on the hematopoietic and immune systems.

Chocolate milk is increasingly recognized as an effective recovery drink due to its optimal carbohydrate-to-protein ratio (approximately 3:1 or 4:1), promoting rapid glycogen replenishment and muscle fiber repair. Studies suggest that post-exercise chocolate milk consumption may be as effective, or even superior, to commercial sports drinks, particularly in endurance recovery. Additionally, chocolate milk provides high-quality milk protein, electrolytes (calcium, potassium, sodium), and lipids, supporting hydration homeostasis and reducing oxidative stress post-exercise. This combination may limit muscle damage, reduce inflammation (lower CK and IL-6 levels), and improve acid-base balance, making chocolate milk a viable nutritional strategy for endurance athletes.

This study aims to evaluate the effectiveness of chocolate milk in kayakers' recovery by analyzing metabolic, inflammatory, and hematological markers, thus determining its potential role in optimizing endurance sports nutrition strategies.

Changes in glucose, glycogen, insulin, CK, IL-6, grhelin, leptin, peptide YY, peripheral blood morphology, and blood gas parameters will be analyzed to better understand recovery and adaptation mechanisms influenced by chocolate milk consumption. Also, the project results may provide a basis for further research on the role of appetite hormones in sports recovery, which is a relatively new area of research in sports dietetics, and have a significant impact on new strategies to support athletes' performance.

Methods This study will examine chocolate milk's effectiveness in 30 elite kayakers (both sexes), split into experimental (n=15, chocolate milk) and control (n=15, water) groups. Blood samples (capillary and venous) will be collected at three time points: before exercise, immediately after exercise, and 1 hour post-consumption.

- Experimental group - up to 30 minutes after the erometer test, consumes 400 ml of chocolate milk.

Control group - up to 30 minutes after the erometer test, consumes 400 ml of water.

- Exercise test: During the preparatory period (April/May), participants will perform an intensive exercise test on a kayak ergometer (Dansprint PRO, Denmark), consisting of covering a distance of 1000 meters in the shortest time possible. The kayak ergometer test will be performed under medical supervision.

* Before the exercise test, a non-invasive anthropometric analysis will be performed using the TANITA MC-780MA body composition analyzer (Tokyo, Japan), to determine body composition: percentage of body fat, body fat mass, lean tissue mass, muscle mass, water and body mass index (BMI).
* Before the ergometer test, a nutrition analysis will be performed using the food diary method.
* Before the exercise test, a meal will be served containing a standardized amount of kcal, protein, fat, carbohydrates and fiber, calculated per kg of the athlete's body weight, in accordance with the nutrition standards for the Polish population edited by Mirosław Jarosz and the recommendations of the International Society of Sports Nutrition.
* During the test, measurements will be taken: travel time, average power, heart rate.

The results will determine whether chocolate milk accelerates energy replenishment, reduces muscle damage, and decreases inflammation compared to water consumption. This research will contribute to optimizing endurance sports nutrition strategies and serve as a basis for further studies on recovery methods.

ELIGIBILITY:
Inclusion Criteria:

* Lack of consent for blood sampling,
* injuries, health issues,
* anti-inflammatory drugs,
* performance-enhancing substances,
* supplements within the last 3 months before the start of the study.

Exclusion Criteria:

* consent to participate in the study,
* regular training regimen,
* current medical examinations,
* no health contraindications.

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Glycogen level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of glycogen [ng/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline Insulin level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption..
  Concentration of insulin [μIU/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline Creatine kinase activity (CK) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concetration of CK [ng/ml]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline interleukin-6 (Il-6) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of Il-6 [pg/mL]. Immunoenzymatic assay method using a diagnostic ELISA Kit
Changes from baseline in lactic acid (LA) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concetration of LA [mmol/l]. Using a portable biochemical photometer Vario Photometer II (Diaglobal, Berlin, Germany) (capillary blood from the ear lobe).
Baseline Appetite Assessment of Athletes Before Exercise Test Using Visual Analogue Scale (VAS). | Day 1: At rest, after the exercise test.
  The Visual Analogue Scale (VAS) measures subjective appetite sensations-linear scale from one to 10 where 10 is the strongest feeling.
Changes from baseline in leptin (LEP) level. | Day 1:At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Satiety regulation marker. Concentration of leptin [pg/ml].ELISA method by the test manufacturer's instructions.
Changes from baseline in peptide YY (PYY) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Satiety regulation marker. Concentration of leptin [pg/ml]. ELISA method by the test manufacturer's instructions.
Changes from baseline in ghrelin (GHRL) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Hunger regulation marker. Concentration of GHRL [pg/ml].ELISA method by the test manufacturer's instructions.
Changes from baseline in acid-base balance - urea nitrogen (BUN) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of BUN [ml/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - anion gap (AGAP) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of AGAP [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - excess base in extracellular fluid (BE ecf) level. | Day1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of Be ecf [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - sodium (Na) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of Na [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - calcium (Ca) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of Ca [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - potassium (K) level | At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of K [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - chlorine (Cl) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of Cl [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - bicarbonate level (cHCO3). | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of cHCO3 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - total plasma CO2 (tCO2) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of tCO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - partial pressure of carbon dioxide (pCO2) | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of pCO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - partial pressure of oxygen (pO2) | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of pO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance -total blood saturation (cSO2) level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of cSO2 [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - urea level. | Day 1:At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of urea [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - crea level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of crea [mg/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - hematocrit [hct] level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of hct [%]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - hemoglobin [chgb] level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of chgb [mmol/l]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).
Changes from baseline in acid-base balance - glucose [glu] level. | Day 1: At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  Concentration of glu [mg/dl]. Using the portable blood gas, electrolyte, and metabolite analyzer (epoc®) (capillary blood from the ear lobe).

SECONDARY OUTCOMES:
Antropometric characteristic - height | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including height (Seca 213 Hamburg, Deutschland) [cm]
Antropometric characteristic - weight | Day 1 after overall fast
  Anthropometric characteristic - weight
Antropometric characteristic - LBM | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including lean body mas (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Antropometric characteristic - TBW | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including total body water (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [kg]
Antropometric characteristic - Water% | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including water (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [%]
Antropometric characteristic - FAT | Day 1 after overall fast
  Prior to the exercise test, we measured the anthropometric parameters, including fat (Tanita BC 418 MA, Tanita Corporation, Tokyo, Japan) [%]
Food record - energy | Day before the Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: energy [kcal]
Food record - protein | Day before the Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: protein [g]
Food record - carobhydrates | Day before the Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: carbohydrates [g]
Food record - fiber | Day before the Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fiber [g]
Food record - fat | Day before the Day 1
  Participants will prepare a food record. The results will be calculated using the dietetykpro program: fat [g]
Peripheral blood morphology | At rest (before the test), directly after the test, and after a 1-hour post-consumption.
  using MYTHIC18 hematology analyzer (Cormay Diagnostics, Geneva, Switzerland). Qualitative and quantitative evaluation of morphological elements of blood (determination in venous blood).

CONTACTS AND LOCATIONS:
Overall Officials: Anna B Kasperska, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznań University of Physical Education, Faculty of Physical Culture in Gorzów Wielkopolski, Gorzów Wielkopolski, Polska, Poland